CLINICAL TRIAL: NCT05773937
Title: A Phase I Clinical Study of the Safety, Tolerability, Pharmacokinetics and Preliminary Antitumor Activity of 9MW2821 in Advanced Malignant Solid Tumors
Brief Title: A Clinical Study of 9MW2821 in Advanced Malignant Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Mabwell (Shanghai) Bioscience Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9MW2821-2021-CP101
Record Dates: First submitted 2023-02-22; First posted 2023-03-17 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Advanced Malignant Solid Tumors

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 9MW2821 (Experimental)
  Interventions: Drug: 9MW2821

INTERVENTIONS:
Drug: 9MW2821 — All subjects will receive a single intravenous (IV) infusion of 9MW2821 once weekly for the first 3 weeks of every 4 week cycle (i.e., on Days 1, 8 and 15).

SUMMARY:
This study is a Phase 1, first-in-human, open-label, dose-escalation and cohort expansion study designed to characterize the safety, tolerability, pharmacokinetics, preliminary antitumor activity and immunogenicity of 9MW2821 administered by intravenous (IV) infusion.

ELIGIBILITY:
Inclusion Criteria:

* Competent to comprehend, sign, and date an independent ethics committee/institutional review board/research ethics board (IEC/IRB/REB) approved informed consent form.
* Male or female subjects aged 18 to 80 years (including 18 and 80 years).
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Phase Ia：Histologically or cytologically confirmed advanced malignant solid tumors (except sarcoma). Phase Ib：Only local advanced or metastatic UC tumors.
* Subjects must have received ICIs or GC/GP therapies in the previous treatment.
* Subjects must submit tumor tissues for test.
* Life expectancy of ≥ 3 months.
* Subjects must have measurable disease according to RECIST (version 1.1).
* Adequate organ functions.
* Sexually active fertile subjects, and their partners, must agree to use methods of contraception during the study and at least 6 months after termination of study therapy.
* Subjects are willing to follow study procedures.

Exclusion Criteria:

* Chemotherapy、radiotherapy or immunotherpy within 14 days prior to the first dose of study drug.
* Preexisting treatment related toxicity Grade ≥ 2 (except alopecia).
* Major surgery within 28 days prior to first dose of study drug.
* History of uncontrolled diabetes mellitus.
* Preexisting peripheral neuropathy Grade ≥ 2.
* Received treatment of ADCs with MMAE payload.
* Any live vaccines within 4 weeks before first dose of study drug or during the study.
* Documented history of clinically significant cardiac or cerebrovascular diseases within 6 months prior to the first dose of study drug.
* Other severe or uncontrolled disease, i.e. severe respiratory system disease, thromboembolic events, active bleeding or active infection.
* Uncontrolled central nervous system metastases.
* History of another malignancy within 3 years before the first dose of study drug. Subjects with curable malignancies are allowed.
* History of autoimmune disease requiring systemic treatment within 2 years before the first dose of study drug.
* Has ocular conditions that may increase the risk of corneal epithelium damage.
* Known sensitivity to any of the ingredients of the investigational product; History of drug abuse or mental illness.
* Any P-glycoprotein (P-gp) inducers/inhibitors or CYP3A4 inducers/inhibitors for high and medium effect within 14 days prior to the first dose of study drug.
* Use of any investigational drug or device within 30 days prior to the first dose of study drug.
* Conditions or situations which may put the subject at significant risk.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-06-21 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events | Up to 28 days post last drug administration

SECONDARY OUTCOMES:
Pharmacokinetic parameter：total antibody (TAb), antibody drug conjugate (ADC), and Monomethyl Auristatin E (MMAE) | 24 months
  Maximum observed concentration (Cmax)
Pharmacokinetic parameter：total antibody (TAb), antibody drug conjugate (ADC), and Monomethyl Auristatin E (MMAE) | 24 months
  Area under the concentration-time curve (AUC)
Pharmacokinetic parameter：total antibody (TAb), antibody drug conjugate (ADC), and Monomethyl Auristatin E (MMAE) | 24 months
  Half-life (t1/2)
Pharmacokinetic parameter：total antibody (TAb), antibody drug conjugate (ADC), and Monomethyl Auristatin E (MMAE) | 24 months
  Clearance (CL)
Objective Response Rate | Up to 24 months
  ORR
Disease Control Rate | Up to 24 months
  DCR
Duration of Response | Up to 24 months
  DoR
Time to Response | Up to 24 months
  TTR
Progression Free Survival | Up to 24 months
  PFS
Overall Survival | Up to 24 months
  OS
Incidence of Anti-Drug Antibody (ADA) | Up to 24 months
  ADA

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Beijing University Cancer Hospital, Beijing, Beijing Municipality

REFERENCES:
- [Derived] Zhou W, Fang P, Yu D, Ren H, You M, Yin L, Mei F, Zhu H, Wang Z, Xu H, Cao Y, Sun X, Xu X, Bi J, Wang J, Ma L, Wang X, Chen L, Zhang Y, Cen X, Zhu X, Lou L, Liu D, Tan X, Yang J, Meng T, Shen J. Preclinical Evaluation of 9MW2821, a Site-Specific Monomethyl Auristatin E-based Antibody-Drug Conjugate for Treatment of Nectin-4-expressing Cancers. Mol Cancer Ther. 2023 Aug 1;22(8):913-925. doi: 10.1158/1535-7163.MCT-22-0743. PMID 37196158